CLINICAL TRIAL: NCT07262034
Title: The Impact of Preoperative Nutritional Intervention on Muscle Mass Preserve in Older Adult Undergoing Elective Surgery: A Prospective Cohort Study (SiPAP Trail) Study
Brief Title: The Impact of Preoperative Nutrition Intervention on Muscle Mass Preserve in Older Adults Undergoing Elective Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Associate Professor, Siriraj Hospital
Other Study IDs: 655/2568 (IRB2)
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Nutrition Status
Keywords: Preoperative; Sarcopenia; Body Composition Analyzer (BIA); Skeletal Muscle Index (SMI)
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcopenia-the progressive loss of muscle mass and strength-is a major clinical issue, especially in surgical patients with malignancy. It's strongly linked to poor postoperative outcomes like increased complications, longer hospital stays, and higher mortality. Surgical stress (trauma, fasting, immobilization) significantly worsens this muscle catabolism.

Consequently, early identification and targeted preoperative intervention are essential. Preoperative nutrition, part of a prehabilitation program, is a key strategy known to attenuate muscle loss and improve recovery. The Skeletal Muscle Index (SMI) is an objective metric used for risk stratification.

The Siriraj Integrated Preoperative and Prehabilitation Center (SiPAP) uses a multidisciplinary model with nutritional counseling, but lacks routine sarcopenia screening or objective SMI measurement. Therefore, the impact of their specific nutritional interventions on preserving muscle mass remains unevaluated.

Hypothesis: The structured, individualized preoperative nutritional intervention delivered by SiPAP to intraabdominal oncology patients will result in a net preservation or positive change in the Skeletal Muscle Index (SMI) over the preoperative period.

DETAILED DESCRIPTION:
Sarcopenia, defined as the progressive loss of skeletal muscle mass and strength, is clinically associated with poor clinical outcomes, increased physical disability, and low quality of life.1 Sarcopenia is common in a geriatric population, but it is also frequently observed in patients with cancer and other chronic conditions..

In patients undergoing surgery, especially those with malignancy, sarcopenia is independently associated with poor postoperative outcomes. It leads to frailty, delayed functional recovery, increased complication rates, prolonged hospital stays, and higher mortality.2-9 For cancer patients, a progressive decrease in muscle mass is a common issue, even during treatment such as neoadjuvant chemotherapy.10-12 This catabolic state is clinically relevant even over short time frames. A reduction of ≥10% in skeletal muscle index is considered clinically meaningful, and even modest short-term losses of 5-10% muscle mass in surgical or oncology patients are associated with poorer clinical outcomes and delayed recovery. 4,6,13-15 The pathophysiology of sarcopenia is multifactorial, involving reduced protein intake, physical inactivity, systemic inflammation, and hormonal changes. Surgical stress exacerbates muscle catabolism through mechanisms such as surgical trauma, perioperative fasting, and postoperative immobilization. 3-6,8,16-19 These effects are particularly concerning in older patients undergoing major procedures.3-6,8,16-19 Consequently, early identification and targeted intervention to preserve muscle integrity are essential of perioperative care for improving postoperative recovery and surgical outcomes. Body composition assessment, particularly using the skeletal muscle index (SMI), is an important metric in preoperative risk stratification and may help identify patients most likely benefit from prehabilitation.

Preoperative nutritional interventions, delivered as part of structured prehabilitation program, represent a key strategy to counteract perioperative muscle wasting. These interventions programs typically involve individualized nutrition counseling, targeted protein supplementation, and physical activity guidance. 20-28 Several studies have demonstrated the beneficial effects of optimizing nutrition to prevent and manage sarcopenia. Tailored dietary advice, with particularly focus on adequate protein intake, has been shown to attenuate muscle mass loss and improve muscle strength in patients at- risk patients of or diagnosed with sarcopenia. 22,24,26,27 In older surgical patients, individualized nutrition interventions are associated with improvements in physical performance measures such as gait speed, and handgrip strength, and short physical performance.27 Furthermore, nutritional guidance, when combined with exercise therapy as part of multimodal prehabilitation, has been reported to enhance muscle protein synthesis, support functional recovery, and reduce sarcopenia progression both before and after surgery. 24,28 These findings highlight the critical role of structured nutritional counseling in preserving skeletal muscle integrity during the perioperative period, aligning with the principles of Enhanced Recovery After Surgery (ERAS) protocols aimed to optimize patients' physical status and accelerating recovery.29-32 The Siriraj Integrated Preoperative and Prehabilitation Center (SiPAP) implements a multidisciplinary prehabilitation model, including comprehensive nutritional counseling and nutritional status assessments, aligned with ERAS principles. However, SiPAP has never formally screened for sarcopenia, nor has it routinely used objective measures of muscle mass, such as Skeletal Muscle Index (SMI) calculated from Bioelectrical Impedance Analysis (BIA). Given the strong association between sarcopenia and poor surgical outcomes, this represents a significant gap in our current risk stratification. Therefore, the impact of the specific, structured preoperative nutritional interventions provided by SiPAP on objective muscle mass preservation (SMI) and the incidence of sarcopenia has not been evaluated in this population.

Therefore, investigators hypothesizes that is that the structured, individualized preoperative nutritional intervention in intraabdominal oncology patients will result in a net preservation or positive change in in skeletal muscle index over the pre-operative period (between the initial SiPAP consultation and hospital admission for elective surgery.

This prospective study aims to determine the absolute mean change in skeletal muscle index (SMI), which will be measured using bioelectrical impedance analysis (BIA) for the first time in this participants cohort, following the nutritional intervention period. Secondary objectives include

1. To quantify the absolute change in body weight (kg) and total calorie and protein intake (kcal/day, g/day) at hospital admission preoperatively.
2. To assess the improvement in nutritional status, defined by a change in PG-SGA, comparing baseline to pre-admission.
3. To establish the baseline prevalence and the change in sarcopenia classification based on AWGS criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 60 years to 90 years
2. Schedules for elective major surgery and formally enrollment in the Enhanced Recovery After Surgery (ERAS) program at Siriraj Hospital. (At Siriraj Hospital, patients scheduled for pre-specific elective major surgeries are enrolled into the ERAS program as individual hospital protocols for each ERAS module. All patients are informed about the ERAS program by their surgical team.)
3. Referred to the SiPAP center for prehabilitation based on established ERAS hospital preoperative protocol.
4. Able to provide written informed consent and willing to undergo all research assessments at both time points.

Exclusion Criteria:

1. Presence of conditions that interfere with bioelectrical impedance analysis (BIA), including an implanted pacemaker or other non-removable electronic medical devices.
2. Use of medications or supplements known to acutely or chronically affect muscle mass (e.g. corticosteroids, hormonal therapies) during the study period.
3. Diagnosed neuromuscular disorders that affect baseline muscle mass and strength
4. Undergo emergency surgery
5. A planned interval of less than 14 days between the initial SiPAP visit and hospital admission for surgery.
6. Alcohol consumption or strenuous exercise within the 12 hours preceding the scheduled BIA measurement.
7. Incomplete data on muscle mass or nutritional assessment at either time point.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who enroll to Enchanced Recovery After Surgery (ERAS) program, Siriraj Hospital and referred to the SiPAP program
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the skeletal muscle index (SMI) at a day admit to surgery | From a preoperative clinic consultation (baseline) to a day admit to surgery, up to 3 months
  Skeletal muscle index (SMI) determined by bioelectrical impedance analysis (BIA) and report as a value with units of kilograms per meter squared (kg/m2)

SECONDARY OUTCOMES:
Change from Baseline in nutrition status at a day admit to surgery | From a preoperative clinic consultation (baseline) to a day admit to surgery, up to 3 months
  Nutrition status defined by Patient-Generated Subjective Global Assessment (PG-SGA).
  The minimum PG-SGA score is 0, while the maximum score is 30. The higher the score, the greater the risk of malnutrition.
Change from Baseline in sarcopenia classification at a day admit to surgery | From a preoperative clinic consultation (baseline) to a day admit to surgery, up to 3 months
  Sarcopenia classification based on the Asian Working Group for Sarcopenia (AWGS) 2019 criteria (Possible Sarcopenia, Sarcopenia, Severe Sarcopenia)
Change from Baseline in the body weight at a day admit to surgery | From a preoperative clinic consultation (baseline) to a day admit to surgery, up to 3 months
  Body weight report as units of kilograms (kg)
Change from Baseline in the total calorie intake at a day admit to surgery | From a preoperative clinic consultation (baseline) to a day admit to surgery, up to 3 months
  Total calorie intake report as units of kcal/day
Change from Baseline in the total protein intake at a day admit to surgery | From a preoperative clinic consultation (baseline) to a day admit to surgery, up to 3 months
  Total protein intake report as units of g/day

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Mingkwan Wongyingsinn, MD, Study Director — Department Of Anesthesiology, Faculty Of Medicine Siriraj Hospital
Locations (1):
- Siriraj Integrated Preoperative And Prehabilitation Center : SiPAP, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chaiwat O, Wongyingsinn M, Muangpaisan W, Chalermsri C, Siriussawakul A, Pramyothin P, Thitisakulchai P, Limpawattana P, Thanakiattiwibun C. A simpler screening tool for sarcopenia in surgical patients. PLoS One. 2021 Sep 23;16(9):e0257672. doi: 10.1371/journal.pone.0257672. eCollection 2021. PMID 34555077
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Nitichai N, Angkatavanich J, Somlaw N, Voravud N, Lertbutsayanukul C. Validation of the Scored Patient-Generated Subjective Global Assessment (PG-SGA) in Thai Setting and Association with Nutritional Parameters in Cancer Patients. Asian Pac J Cancer Prev. 2019 Apr 29;20(4):1249-1255. doi: 10.31557/APJCP.2019.20.4.1249. PMID 31030501
- [Background] Taylor BE, McClave SA, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society of Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). Crit Care Med. 2016 Feb;44(2):390-438. doi: 10.1097/CCM.0000000000001525. No abstract available. PMID 26771786
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Arribas L, Sabate-Llobera A, Domingo MC, Taberna M, Sospedra M, Martin L, Gonzalez-Tampan AR, Pallares N, Mesia R, Baracos VE. Assessing dynamic change in muscle during treatment of patients with cancer: Precision testing standards. Clin Nutr. 2022 May;41(5):1059-1065. doi: 10.1016/j.clnu.2022.03.016. Epub 2022 Mar 11. PMID 35395556